CLINICAL TRIAL: NCT04292262
Title: A Prospective Observational Study on the Incidence of Acute Kidney Injury in Polytrauma Patients in Intensive Care Unit
Brief Title: Acute Kidney Injury in Polytrauma Patients in Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Abdallah ElGendy MD, Assistant Professor, Ain Shams University
Other Study IDs: FMASU M S 289/2020
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: AKI (Acute Kidney Injury) Due to Trauma
MeSH Terms: conditions — Acute Kidney Injury | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI
  Interventions: Other: Observational
- Non AKI
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
Acute Kidney Injury (AKI) is a common complication of severe trauma patients and is associated with increased morbidity and mortality.Trauma patients have many risk factors for AKI such as hypovolemic shock, rhabdomyolysis, massive transfusion, major surgeries and abdominal compartment syndrome.The primary outcome of the study is to correlate between the AKI by using RIFLE criteria and the trauma severity by using ISS .The secondary outcomes are ;the length of ICU and hospital stay and 28 days mortality in AKI patients.

DETAILED DESCRIPTION:
• Study Population: 60 cases of polytrauma patients who have ISS>15.

* Inclusion Criteria:

  * Age from 18 to 70 years old males or females
  * Injury Sensitivity Score (ISS >15 )
* Exclusion Criteria:

Patients have end stage liver disease, end stage kidney disease, disseminated malignancy or decompensated heart failure.

Sample size :the calculated sample size is 60 cases of trauma patients.

• All patients' data will be recorded on admission and daily for 7 days:

* Vital signs (blood pressure, heart rate, respiratory rate, body temperature).
* Lab investigations: complete blood count, international normalized ratio, prothrombin time, arterial blood gases, kidney function tests, liver function tests, creatine kinase, creatine kinase-muscle band, creatinine clearance, serum sodium, serum potassium and serum phosphorus will be requested for all patients at admission then daily follow up by creatine kinase, creatine kinase-muscle band, kidney function tests, serum sodium, serum potassium and serum phosphorus for 7 days. Glasgow Coma Scale (GCS), Injury Severity Score (ISS),Urine output (ml/kg/h),RIFLE criteria.,Length of ICU and hospital stay,28 days mortality.

ELIGIBILITY:
Inclusion Criteria:

* • Age from 18 to 70 years old males or females

  * Injury Sensitivity Score (ISS >15 )

Exclusion Criteria:

* Patients have end stage liver disease, end stage kidney disease, disseminated malignancy or decompensated heart failure.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: a prospective observational cohort study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Correlate between the AKI by using RIFLE criteria and the trauma severity by using ISS | 7 days

SECONDARY OUTCOMES:
the length of ICU and hospital stay and 28 days mortality in AKI patients. | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa El Gendy, Cairo, Ain Shams University Specialized Hospital, Egypt

IPD SHARING:
Plan to Share IPD: No